CLINICAL TRIAL: NCT02403986
Title: A Randomised, Multi-centre, Parallel-group, Efficacy and Safety Study Evaluating Two and Three Initial Treatment Sessions of Restylane Skinboosters Vital Lidocaine in the Face
Brief Title: An Efficacy and Safety Study Evaluating Treatment Sessions of Restylane Skinboosters Vital Lidocaine in the Face
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CTN 05DF1404
Record Dates: First submitted 2015-03-26; First posted 2015-03-31 (Estimated); Results first posted 2019-09-06 (Actual); Last update posted 2022-08-26 (Actual); Status verified 2019-09

CONDITIONS: Aged Skin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- R. Vital Skinboosters Lidocaine (three) (Experimental): Treatment with three initial sessions
  Interventions: Device: Restylane Vital Skinboosters Lidocaine
- R. Vital Skinboosters Lidocaine (two) (Experimental): Treatment with two initial sessions
  Interventions: Device: Restylane Vital Skinboosters Lidocaine

INTERVENTIONS:
Device: Restylane Vital Skinboosters Lidocaine

SUMMARY:
A randomised, multi-centre, parallel-group efficacy and safety study evaluating two and three initial treatment sessions of Restylane Skinboosters Vital Lidocaine in the face.

DETAILED DESCRIPTION:
Approximately 50 female subjects shall be treated with two or three initial treatment sessions including long-term follow-up 18 months after the initial treatment regimen. Efficacy and safety to be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent to participate in the study.
* Non-pregnant, non-breast feeding female aged 35-45 years.
* Visible signs of aging in the face
* Intent to improve skin hydration, skin structure and the elasticity of the skin using - Restylane Skinboosters Vital Lidocaine.

Exclusion Criteria:

* Extensively photo damaged and aged skin.
* Woman who plan to become pregnant during the course of the study.
* Known/previous allergy or hypersensitivity to any injectable hyaluronic acid (HA) gel.
* Known/previous allergy or hypersensitivity to local anaesthetics, e.g. lidocaine or other amide-type anaesthetics.
* History of severe or multiple allergies manifested by anaphylaxis.
* History of bleeding disorders or treatment with anticoagulants or inhibitors of platelet aggregation, Omega-3 or Vitamin E within 10 days before study treatment
* Treatment with chemotherapy, immunosuppressive agents, immunomodulatory therapy (e.g. monoclonal antibodies), systemic or topical (facial) corticosteroids (inhaled corticoids are allowed) within three months before study treatment.
* Previous tissue augmenting therapy or contouring with permanent filler or fat-injection in the face.
* Previous tissue augmenting therapy, contouring or revitalisation treatment with non-permanent filler, neurotoxin or revitalisation preparations (e.g. Hyal System or Restylane Skinboosters) in the face within 12 months before study treatment.
* Previous tissue revitalisation treatment with laser or light, radiofrequency, focused ultrasound, chemical peeling, dermabrasion, mesotherapy or any other similar treatment with influence on skin quality in the face within 6 months before study treatment.
* Previous aesthetic facial surgical therapy, liposuction or tattoo in the face.
* Previous sinus surgery or dental root surgery within 3 months before study treatment.
* Active skin disease, inflammation or related conditions, such as infection, perioral dermatitis, seborrheic eczema, rosacea, acne, psoriasis or herpes zoster in the face.
* History of or active collagen diseases or autoimmune diseases such as systemic lupus erythematosus, rheumatic arthritis, skin or systemic sclerosis.
* Tendency to form keloids, hypertrophic scars or any other healing disorder.
* History of radiation of or cancerous or pre-cancerous lesions (e.g. actinic keratosis) in the face.
* Use of systemic or facial topical retinoic acid within 12 months before study treatment.
* Nicotine use within 6 months before study treatment. (Occasional smoking, such as 1-5 cigarettes per week, or similar amount of nicotine, is allowed).
* Any medical condition that, in the opinion of the Investigator, would make the subject unsuitable for inclusion (e.g. chronic, relapsing or hereditary disease that may interfere with the outcome of the study.
* Other condition preventing the subject from entering the study in the Investigator's opinion, e.g. subjects not likely to avoid other facial aesthetic treatments, subjects anticipated to be unreliable, unavailable or incapable of understanding the study assessments or having unrealistic expectations of the treatment result.
* Study site personnel or close relatives of the study site personnel (e.g. parents, children, siblings and spouse) or employees at the Sponsor company.
* Participation in any other clinical study within 3 months before study treatment.

Ages: 35 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 53 (Actual)
Dates: Start 2015-04; Primary Completion 2017-03-30 (Actual); Study Completion 2017-03-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gerhard Sattler, MD, Principal Investigator — Rosenpark Research; Martina Kerscher, MD, Principal Investigator — University of Hamburg-Eppendorf
Locations (1):
- Rosenpark Research, Darmstadt, Germany

RESULTS

PARTICIPANT FLOW:
Groups:
- R. Vital Skinboosters Lidocaine (Three): Treatment with three initial sessions
  Restylane Vital Skinboosters Lidocaine
- R. Vital Skinboosters Lidocaine (Two): Treatment with two initial sessions
  Restylane Vital Skinboosters Lidocaine
Period: Overall Study
Arm/Group | R. Vital Skinboosters Lidocaine (Three) | R. Vital Skinboosters Lidocaine (Two)
Started | 26 | 27
Completed | 21 | 23
Not Completed | 5 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | R. Vital Skinboosters Lidocaine (Three) | R. Vital Skinboosters Lidocaine (Two) | Total
Number analyzed (Participants) | 26 | 27 | 53
Age, Continuous [Mean (Full Range); unit: years] | 41.2 [35 to 46] | 41.0 [34 to 46] | 41.1 [34 to 46]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 27 | 53
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 26 | 26 | 52
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Germany | 26 | 27 | 53

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Improved Participants on the Global Aesthetic Improvement Scale (GAIS)-Subject
Description: Subject assessment at follow-up visits of aesthetic change from baseline of the treated areas using the Global Aesthetic Improvement Scale (GAIS).
  GAIS is a 5-graded scale: worse; no change; improved; much improved; or very much improved.
  A clinically significant improvement was defined as a score of improved; much improved; or very much improved.
Time Frame: Baseline, 1 Month, 3 Months, 6 Months, 9 Months, 12 Months, 15 Months, 18 Months
Population: At 1 Month after initial treatment, there were 24 participants in Group A and 25 participants in Group B. (26 and 27 respectively randomized, as reported in Participant Flow.)
Measure: Number (95% Confidence Interval); unit: % improved participants
Arm/Group | R. Vital Skinboosters Lidocaine (Three) | R. Vital Skinboosters Lidocaine (Two)
Number analyzed (Participants) | 24 | 25
% improved participants
  1 month | 91.7 [73.0 to 99.0] | 80.0 [59.3 to 93.2]
  3 months | 79.2 [57.8 to 92.9] | 72.0 [50.6 to 87.9]
  6 months: number analyzed (Participants) | 23 | 24
  6 months | 78.3 [56.3 to 92.5] | 58.3 [36.6 to 77.9]
  9 months: number analyzed (Participants) | 22 | 24
  9 months | 77.3 [54.6 to 92.2] | 50.0 [29.1 to 70.9]
  12 months: number analyzed (Participants) | 22 | 23
  12 months | 81.8 [58.1 to 94.6] | 60.9 [38.5 to 80.3]
  15 months: number analyzed (Participants) | 21 | 22
  15 months | 81.0 [58.1 to 94.6] | 68.2 [45.1 to 86.1]
  18 months: number analyzed (Participants) | 21 | 22
  18 months | 81.0 [58.1 to 94.6] | 77.3 [54.6 to 92.2]

2. Primary Outcome: Percentage of Improved Participants on the Global Aesthetic Improvement Scale (GAIS)-Investigator
Description: Investigator assessment at follow-up visits of aesthetic change from baseline of the treated areas using the Global Aesthetic Improvement Scale (GAIS).
  GAIS is a 5-graded scale: worse; no change; improved; much improved; or very much improved.
  A clinically significant improvement was defined as a score of improved; much improved; or very much improved.
Time Frame: Baseline, 1 Month, 3 Months, 6 Months, 9 Months, 12 Months, 15 Months, 18 Months
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: % improved participants
Arm/Group | R. Vital Skinboosters Lidocaine (Three) | R. Vital Skinboosters Lidocaine (Two)
Number analyzed (Participants) | 24 | 25
% improved participants
  1 month | 100.0 [85.8 to 100.0] | 96.0 [79.6 to 99.9]
  3 months | 95.8 [78.9 to 99.9] | 92.0 [74.0 to 99.0]
  6 months: number analyzed (Participants) | 23 | 24
  6 months | 82.6 [61.2 to 95.0] | 87.5 [67.6 to 97.3]
  9 months: number analyzed (Participants) | 22 | 24
  9 months | 81.8 [59.7 to 94.8] | 70.8 [48.9 to 87.4]
  12 months: number analyzed (Participants) | 22 | 23
  12 months | 86.4 [65.1 to 97.1] | 87.0 [66.4 to 97.2]
  15 months: number analyzed (Participants) | 21 | 22
  15 months | 95.2 [76.2 to 99.9] | 95.5 [77.2 to 99.9]
  18 months: number analyzed (Participants) | 21 | 22
  18 months | 100.0 [83.9 to 100.0] | 90.9 [70.8 to 98.9]

ADVERSE EVENTS:
Time Frame: 18 months
Arm/Group | R. Vital Skinboosters Lidocaine (Three) | R. Vital Skinboosters Lidocaine (Two)
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/27
Serious Adverse Events (participants affected / at risk) | 2/26 | 1/27
Other Adverse Events (participants affected / at risk) | 13/26 | 10/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | R. Vital Skinboosters Lidocaine (Three) (N=26) | R. Vital Skinboosters Lidocaine (Two) (N=27)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Face oedema (General disorders) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | R. Vital Skinboosters Lidocaine (Three) (N=26) | R. Vital Skinboosters Lidocaine (Two) (N=27)
Influenza (Infections and infestations) | 4 (5) | 3 (3)
Viral upper respiratory tract infection (Infections and infestations) | 8 (12) | 5 (7)
Headache (Nervous system disorders) | 2 (2) | 0 (0)
Menopausal symptoms (Reproductive system and breast disorders) | 2 (2) | 0 (0)
Implant site swelling (General disorders) | 2 (5) | 2 (6)
Implant site nodule (General disorders) | 0 (0) | 2 (3)
Implant site pain (General disorders) | 0 (0) | 2 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-12-02): https://cdn.clinicaltrials.gov/large-docs/86/NCT02403986/Prot_SAP_000.pdf